CLINICAL TRIAL: NCT07351188
Title: Survey of Our Healthcare Professionals and Future Healthcare Professionals on Their Training, Knowledge, and Experience Regarding Organ Donation
Brief Title: Survey of Our Future Healthcare Professionals on Their Training, Knowledge, and Experience Regarding Organ Donation
Acronym: Info-PMO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9949
Record Dates: First submitted 2026-01-09; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Organ Donation
Keywords: Organ Donation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2024, 29,000 people were waiting for an organ transplant in France, and only 6,034 transplants were performed during the year. 852 people died in 2024 while waiting for a transplant. The gap between the number of available transplants and the number of patients waiting for a transplant has been widening since the 1990s; there is talk of a shortage of transplants. There is therefore an urgent need to find more transplants and mobilize the entire population to this end.

There are many prejudices and misconceptions about organ donation, which hinder its acceptance. In fact, the rate of opposition to donation has only increased in recent years. Even among the healthcare community, organ donation suffers from a lack of knowledge, which potentially contributes to difficulties in acceptance. This lack of knowledge is probably linked to insufficient training and practice.

The aim of the research is to study the perception of training, knowledge, and experience of organ donation by our healthcare professionals and future healthcare professionals in Alsace, France.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals currently working in a hospital in Alsace, France: state-certified nurse anesthetists, state-certified operating room nurses and operating room nurses, nursing assistants, midwives, dentists, physical therapists, doctors
* Future healthcare professionals currently in training in Alsace: medical/health students, state-certified nurse anesthetist students, operating room nurse students, nursing assistant students, midwife students, dentist students, physical therapist students

Exclusion Criteria:

* Healthcare professionals or future healthcare professionals practicing outside Alsace

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - Healthcare professionals and future healthcare professionals currently training in Alsace:
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03-27 (Estimated)

PRIMARY OUTCOMES:
Percentage of responses: Sufficient, Clear, Useful | Up to 12 months
  This study seeks to understand what healthcare professionals and students in Alsace think about the training they receive on organ donation, to determine if it is sufficient, clear, and useful.
  Percentage of responses: Sufficient, Clear and Useful

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie, Réanimation et Médecine Périopératoire - CHU de Strasbourg - France, Strasbourg, France